CLINICAL TRIAL: NCT06443541
Title: SCALE: Strategies for Implementing GlobalConsent to Prevent Sexual Violence in University Men
Brief Title: Strategies for Implementing GlobalConsent to Prevent Sexual Violence in University Men
Acronym: SCALE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH); Center for Creative Initiatives in Health and Population (Other); Georgia State University (Other)
Responsible Party: Principal Investigator, Kathryn Yount, Professor of Global Health, Emory University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: STUDY00006481; 1R01MH133259 (NIH)
Record Dates: First submitted 2024-05-15; First posted 2024-06-05 (Actual); Last update posted 2025-08-05 (Actual); Status verified 2025-07

CONDITIONS: Violence, Sexual
Keywords: Behavioral Intervention; GlobalConsent; Sexual Violence
MeSH Terms: conditions — Coitus

STUDY DESIGN:
Intervention Model Description: This cluster-randomized design assigns seven universities to High-intensity implementation strategies (HIS) or Lower-intensity (LIS) implementation strategies to deliver GlobalConsent education.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Students (Experimental): Students in either randomization group will become active consumers of GlobalConsent with an email introduction to the program, process, delivery schedule, data collection procedures, and consent.
  Interventions: Behavioral: High-intensity implementation strategies (HIS)-Students; Behavioral: Low-intensity implementation strategies (LIS) for Students
- Faculty (Experimental): Faculty will receive access to educational material based on the university randomization implementation strategies group.
  Interventions: Other: High-intensity implementation strategies (HIS) for Faculty; Other: Low-intensity implementation strategies (LIS) for Faculty
- Leaders (Experimental): Leaders will receive site-specific (University) invitations and material based on the implementation strategies group.
  Interventions: Other: High-intensity implementation strategies (HIS) for Leaders; Other: Low-intensity implementation strategies (LIS) for Leaders
- Implementation Team Members (Experimental): Implementation team members will receive passive access to web-based materials and training according to the university-specific implementation strategies group.
  Interventions: Other: High-intensity implementation strategies (HIS) for Implementation Team Members; Other: Low-intensity implementation strategies (LIS) Implementation Team Members

INTERVENTIONS:
Behavioral: High-intensity implementation strategies (HIS)-Students — Students in the HIS group will receive educational outreach in a pre-implementation in-person orientation to GlobalConsent, covering similar topics and three monthly one-hour learning sessions during implementation in which technical questions about program access or progression can be addressed; more intensive intervention to enhance adherence with more frequent email/Short Message Service (SMS), completion reminders; and demand generation encouraging program completion.
  Other Names: HIS-Students
  Arms: Students
Behavioral: Low-intensity implementation strategies (LIS) for Students — Students in the LIS group will receive basic implementation strategies of the GlobalConsent often used to deliver online programs at US universities with email/SMS completion reminders with a predetermined frequency for 12 weeks.
  Other Names: LIS-Students
  Arms: Students
Other: High-intensity implementation strategies (HIS) for Faculty — * Passive access to web-based educational materials
  * Town halls (3) with general faculty to define sexual violence; rates in young people; acute/chronic effects over the life course; primary-prevention evidence-based interventions (EBIs)
  Other Names: HIS-Faculty
  Arms: Faculty
Other: Low-intensity implementation strategies (LIS) for Faculty — Passive access to web-based educational materials
  Other Names: LIS-Faculty
  Arms: Faculty
Other: High-intensity implementation strategies (HIS) for Leaders — * Site-specific invitation to participate
  * Passive access to web-based educational materials
  * One pre-implementation webinar to define sexual violence; rates among young people in Vietnam; acute/chronic effects over life course; primary-prevention EBIs; recap of project description and collaboration; share GlobalConsent website for passive access to educational materials
  * Monthly emails from trained internal facilitators to university leaders with updates on implementation progress
  * One post-implementation webinar to share anonymized findings (by IS group); discuss plan for sustainment (including guidance on how to handle reporting of sexual violence in existing university counseling centers)
  Other Names: HIS-Leaders
  Arms: Leaders
Other: Low-intensity implementation strategies (LIS) for Leaders — * Site-specific invitation to participate
  * Passive access to web-based educational materials
  * One pre-implementation webinar to define sexual violence; rates among young people in Vietnam; acute/chronic effects over life course; primary-prevention EBIs; recap of project description and collaboration; share GlobalConsent website for passive access to educational materials
  Other Names: LIS-Leaders
  Arms: Leaders
Other: High-intensity implementation strategies (HIS) for Implementation Team Members — * Passive access to web-based educational materials
  * In-person technical training on campus-wide implementation of GlobalConsent; discussion and demonstration of GlobalConsent program; standardized implementation manual
  * In-person leadership training to champion GlobalConsent with internal stakeholders (leaders, implementation teams, faculty, students); leadership styles; managing teams; influence without authority; managing conflict; emotional intelligence; negotiation; leading change
  * Biweekly (six) 1-hr recorded quality-improvement team webinars to provide refresher training; assess implementation progress; assess modifications; build peer-network; provide anonymized data on implementation progress for discussion
  Other Names: HIS-Implementation Team Members
  Arms: Implementation Team Members
Other: Low-intensity implementation strategies (LIS) Implementation Team Members — * Passive access to web-based educational materials
  * In-person technical training on campus-wide implementation of GlobalConsent; discussion and demonstration of GlobalConsent program; standardized implementation manual
  Other Names: LIS Implementation Team Members
  Arms: Implementation Team Members

SUMMARY:
This project, SCALE, will be the first to compare lower-intensity (standard) and higher-intensity implementation strategies to deliver GlobalConsent-an efficacious web-based sexual violence prevention program-to men attending seven universities across Vietnam. Following a rigorous, mixed-methods, comparative interrupted-time-series design, researchers will collect novel data to compare implementation fidelity, drivers and outcomes, effectiveness, and cost-effectiveness across implementation strategy groups. This partnership includes universities also engaged in a violence-prevention training grant (D43TW012188), offering an unparalleled opportunity for capacity strengthening and evidence generation to guide national leaders on the best strategies for launching GlobalConsent at scale, addressing a sex-differentiated risk factor in adolescence, and thereby improving a range of health outcomes into adulthood.

DETAILED DESCRIPTION:
Sexual violence is prevalent in adolescence and heightens the risk of harmful long-term health effects. Sexual violence includes any sexual act committed against a person without freely given consent. All sexes may experience sexual violence, but sexual violence more often burdens women than men globally, and men most often perpetrate such violence. Adolescence is a period of vulnerability to sexual violence, with about one in five college women in the US experiencing a campus sexual assault, and 91% of victims being women. Less is known about the rates of sexual violence on college campuses. Still, estimates from large, multi-country surveys confirm that young men's reported sexually violent behavior and young women's reported sexual violence victimization are high, including in Asia/Pacific. In Vietnam, from 2010 to 2019, women's reports of lifetime sexual violence by a partner increased (10% to 13%), especially in women 18-24 years (5% to 14%). Such trends may reflect changing exposure and more openness to discuss sex and sexual violence. Also, nearly one in ten women (9%) report non-partner sexual violence since age 15, mostly perpetrated by non-family male acquaintances, co-workers, or strangers. Young women who are victims of sexual violence are at heightened risk of acute and chronic mental and physical health conditions.

The researchers will use the Reach, Effectiveness, Adoption, Implementation, and Maintenance (RE-AIM) and Proctor et al. frameworks and a mixed-methods, comparative interrupted time series (CITS) design to compare implementation; implementation drivers and outcomes; implementation effectiveness; and cost-effectiveness of lower-intensity vs higher-intensity (LIS; HIS) implementation strategies to deliver GlobalConsent.

ELIGIBILITY:
Inclusion Criteria for Students:

* 18 and older
* Men who self-identify as heterosexual or bisexual (who are attracted to women),
* Enrolled as first-year students in any of the seven participating study universities in North, Central, and South Vietnam.

Exclusion Criteria for Students:

* Adults unable to consent
* Individuals who are not yet adults (infants, children, teenagers)

Inclusion Criteria for Faculty:

* All registered lecturers at each of the seven participating study universities will be eligible to participate in the faculty surveys in years 1, 3, and 5.

Exclusion Criteria for Faculty:

* None

Inclusion Criteria for Leaders:

* Recommendation of study staff at each participating study university
* Knowledge about the implementation landscape and implementation of GlobalConsent.

Exclusion Criteria for Leaders:

* None

Inclusion Criteria for Implementation Teams:

* Identified by relevant study staff.

Exclusion Criteria for Implementation Teams:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 3439 (Estimated)
Dates: Start 2024-03-27 (Actual); Primary Completion 2028-02 (Estimated); Study Completion 2028-02 (Estimated)

PRIMARY OUTCOMES:
Students' Reported Prosocial Bystander Behavior | Baseline, every 6 months up to 30 months
  Students will be asked if they had engaged in any of seven prosocial bystander behaviors in the past 3 months (or since the last time completing the questionnaire). Items are scored as 0 = never performed, 1 = performed once, 2 = performed more than once. The numbers of participants who report engaging in at least one of seven prosocial bystander behaviors at least once are presented here.
Students' reported Sexually Violent Behavior | Baseline, every 6 months up to 30 months
  The Sexual Experiences Survey (SES) is an assessment tool used to measure the prevalence of sexual aggression. It is designed to measure the frequency and severity of sexual aggression acts committed by an individual. The SES is a self-report questionnaire developed by researchers at the University of Michigan. The Sexual Experiences Survey - Short Form Victimization is a multi-item measure to assess unwanted sexual victimization. Surveys will be provided every six months for up to 30 months.

SECONDARY OUTCOMES:
Perceptions of Sexual Violence form at their respective university | Baseline and up to 49 months
  Perceptions of sexual violence will be assessed by respondents rating their level of agreement with 3 statements regarding the frequency and impact of sexual violence at their university using a 5-point Likert scale ranging from "Totally disagree" to "Totally agree."
  Surveys will be provided to all groups at different time points as below:
  * Students: Baseline, every 6 months up to 30 months
  * Faculty: Baseline, 24 months, and 49 months
  * Leaders: Baseline and 36 months
  * Implementation Team: Baseline, month 15, month 18, and month 42
Implementation Team Scale for staff and supervisors | Baseline, month 15, month 18, and month 42
  Leadership in implementation teams is assessed using two scales, one for implementation team supervisors, and one for implementation team staff. Each scale has 13 items and uses a 5-point Likert ranging from "Totally disagree" to "Totally agree" to assess respondent's agreement on statements about their team supervisor (for staff) or themselves (for supervisors).
Cultural Exchange Inventory | Baseline, month 15, month 18, and month 42
  For implementation team members only: The Cultural Exchange Inventory assesses the teamwork landscape of GlobalConsent implementation teams using 7 items. Respondents give their level of agreement, using a 5-point Likert scale ranging from "Totally disagree" to "Totally agree," on statements such as "The implementation team is working well together to implement GlobalConsent" and "My colleagues are devoting a lot of time and energy to maintain the collaboration of the implementation team.
College Date Rape Attitudes & Behaviors Scale | Baseline, month 15, month 18, and month 42
  For implementation team members only: The College Date Rape Attitude Survey (CDRAS), a measure intended to assess attitudes related to the risk of committing rape in adolescents and young adults, the CDRAS measures four rape-related attitudes: Entitlement, Blame Shifting, Traditional Roles, and Overwhelming Sexual Arousal. The CDRAS contains 20 items measuring attitudes toward date rape. All items require responses on a 5-point Likert scale. The responses for the attitude scale are strongly agree, agree, neutral, disagree, and strongly disagree. Scoring is reversed for appropriate items; so that high scores (5) always correspond to the most desirable (rape-related) responses.
Acceptability, Feasibility, and Appropriateness of Programming to Prevent Sexually Violent Behavior among Students | Baseline and up to 49 months
  This scale assesses respondents' attitudes towards sexual violence prevention programming by asking them to rate their level of agreement with 10 statements, such as "Implementing sexual violence prevention programming with students at our university is something I support," "...addresses a relevant problem among our students," "…would be easy for students to participate in." These statements will be rated using a 5-point Likert scale ranging from "Totally disagree" to "Totally agree."
  Surveys will be provided to all groups at different time points as below:
  * Students: Baseline, every 6 months up to 30 months
  * Faculty: Baseline, 24 months, and 49 months
  * Leaders: Baseline and 36 months
  * Implementation Team: Baseline, month 15, month 18, and month 42
Acceptability, Feasibility, and Appropriateness of GlobalConsent | Baseline and up to 49 months
  This scale assesses respondents' attitudes towards the GlobalConsent program specifically by asking them to rate their level of agreement or disagreement with 10 statements, such as "Implementing GlobalConsent with students at our university is something I support," "...addresses a relevant problem among our students," "…would be easy for students to participate in." these statements will be rated using a 5-point Likert ranging from "Totally disagree" to "Totally agree."
  Surveys will be provided to all groups at different time points as below:
  * Students: Baseline, every 6 months up to 30 months.
  * Faculty: Baseline, 24 months, and 49 months
  * Leaders: Baseline and 36 months
  * Implementation Team: Baseline, month 15, month 18, and month 42
Sexual Violence Legality and Harm (Information about Sexual Activity) | Baseline and up to 49 months
  Knowledge of the law is assessed with 12 items where respondents indicate if they think the situations described are illegal (scored as 1), legal, but harmful (2), or legal and not harmful (3), with example items including "Forcing a person to have oral sex" and "Pressuring someone to have sex." Items will be re-coded such that responses indicating an accurate estimate or overestimate of the illegality and harms of sexual violence were coded as "1" and items indicating an underestimation of the illegality and harms of sexual violence were coded as "0".
  Surveys will be provided to all groups at different time points as below:
  * Students: Baseline, every 6 months up to 30 months.
  * Faculty: Baseline, 24 months, and 49 months
  * Leaders: Baseline and 36 months
  * Implementation Team: Baseline, month 15, month 18, and month 42
Active Consent (Information about Sexual Consent) | Baseline and up to 49 months
  This form adapted the Sexual Consent Scale to ask respondents to rate their level of agreement with 12 statements about sexual consent using a 5-point Likert scale ranging from "totally disagree" to "totally agree". It includes statements such as "If a person consents to sex, one can continue sexual contact even if the person changes their mind," and "Obtaining consent for sex is just as necessary in a long-term relationship as in a new relationship."
  Surveys will be provided to all groups at different time points as below:
  * Students: Baseline, every 6 months up to 30 months
  * Faculty: Baseline, 24 months, and 49 months
  * Leaders: Baseline and 36 months
  * Implementation Team: Baseline, month 15, month 18, and month 42
Rejection of Rape Myths (Attitudes about Sexual Situations) | Baseline and up to 49 months
  This form is a combination of the Illinois Rape Myth Acceptance Scale and the College Date Rape Attitudes & Behaviors Scale. This assesses attitudes towards sexual assault and rape by asking respondents to rate their level of agreement or disagreement with 15 statements using a 5-point Likert ranging from "totally disagree" to "totally agree". Statements include "If a woman dresses in a sexy dress, she is asking for sex," and "When guys rape, it is usually because of their strong desire for sex."
  Surveys will be provided to all groups at different time points as below:
  * Students: Baseline, every 6 months up to 30 months.
  * Faculty: Baseline, 24 months, and 49 months
  * Leaders: Baseline and 36 months
  * Implementation Team: Baseline, month 15, month 18, and month 42
Perceptions of Campus Attittudes | Baseline and up to 49 months
  This form assesses the perceptions of respondents in their university's faculty and leaders' potential response to sexual violence on their university campus. Questions ask about behaviors of abuse, sexual assault, and stalking, and their level of agreement or disagreement with whether faculty and leaders would believe a student reporting experiencing these behaviors, respect a student who reported experiencing these behaviors, or admire a student intervening in these behaviors. Agreement is assessed using a 5-point Likert scale ranging from "totally disagree" to "totally agree"
  Surveys will be provided to all groups at different time points as below:
  * Students: Baseline, every 6 months up to 30 months
  * Faculty: Baseline, 24 months, and 49 months
  * Leaders: Baseline and 36 months
  * Implementation Team: Baseline, month 15, month 18, and month 42
Alcohol Impairment Knowledge/Effects of Alcohol on Cognition | Baseline, every 6 months for up to 30 months.
  Students only: This form asks respondents' agreement or disagreement on 5 alcohol-related questions focusing on decision-making, behavior, and sexual violence. It assesses agreement or disagreement using a 5-point Likert ranging from "totally disagree" to "totally agree".
Empathy for Rape Victims | Baseline, every 6 months for up to 30 months.
  Students only: Empathy for rape victims will be assessed with a modified version of the Rape Empathy Scale (RES). This assessment includes 10 items where participants were asked to choose between two statements, one of which reflected greater empathy towards rapists ("I understand the helplessness a rapist might feel during a rape since he cannot control his actions") and one of which reflected greater empathy towards victims ("I understand the helplessness a victim might feel during a rape"). Responses are scored as 1 (more empathy for victim) or 0 (more empathy for perpetrator) and total scores range from 0 to 10 where higher scores indicate more empathy towards rape victims.
Sexual Communication Attitudes | Baseline, every 6 months for up to 30 months.
  Students only: This is a 7-item scale measuring agreement or disagreement with statements focusing on sexual communication. Agreement and disagreement is assessed using a 5-point Likert ranging from "totally disagree" to "totally agree."
Bystander Self-Efficacy | Baseline, every 6 months for up to 30 months.
  Students only: Bystander Self-Efficacy will be measured using the Bystander Efficacy Scale, which was developed for a project that evaluated the effectiveness of a sexual violence prevention program based on preventing antecedents to sexual violence by increasing prosocial bystander behavior. On this measure, participants are asked to indicate their confidence, on a 3-point scale, in performing each of 10 bystander behaviors (e.g., "Speak up to a guy who is making excuses for using physical force in a sexual relationship."). Scores are created by subtracting the mean of the 10 items from 100 to create a scale of perceived ineffectiveness; thus, higher scores indicate lesser effectiveness.
Bystander Intention to Intervene (Readiness to Intervene) | Baseline, every 6 months for up to 30 months.
  Students only: Readiness to Intervene will be measured using three intent-to-help subscales.
  * Intent to Help Friend Scale: Sexual Abuse
  * Intent to Help Friend Scale: Intimate Partner Violence Intent to help is an attitude that is related to bystander action. Participants will be asked how likely they are to take different bystander actions.
  The second Intent to Help subscale focuses on participants' intent to help strangers in both sexual abuse and intimate partner abuse situations.
  Responses range from 1 (not at all likely) to 5 (extremely likely). The average is calculated from the answers across the items to score this measure.
Severity Measure for Depression | Baseline
  Students only: Depression will be measured using the Patient Health Questionnaire 9 (PHQ-9): The PHQ-9 is a multipurpose instrument for screening, diagnosing, monitoring, and measuring the severity of depression. The PHQ-9 is completed by the participant in minutes and is rapidly scored by a clinician. The PHQ-9 can also be administered repeatedly, which can reflect the improvement or the worsening of depression in response to treatment. PHQ-9 scores of 5, 10, 15, and 20 represent mild, moderate, moderately severe, and severe depression.
Generalized Anxiety Disorder | Baseline
  Students will complete the Generalized Anxiety Disorder 7-item (GAD-7), which is a quick and easy tool to help identify patients with anxiety and monitor treatment response. The GAD-7 has been validated as a diagnostic tool and a severity assessment scale. The scale consists of 7 items. The total score can range from 0 to 21, and it indicates the severity of anxiety as follows:
  0 to 4: Minimal anxiety 5 to 9: Mild anxiety 10 to 14: Moderate anxiety 15 to 21: Severe anxiety
Disability Assessment and Schedule | Baseline
  Students only: The Disability Assessment will be assessed by using the World Health Organization Disability Assessment Schedule 2.0 (WHODAS 2.0), which is a generic assessment instrument for health and disability used across all diseases, including mental, neurological and addictive disorders, applicable in both clinical and general population settings. It is a tool to measure the level of disability and functioning in six domains. The answers rate each question on a scale from 0 (none) to 4 (extreme or cannot do).
  There are three scoring methods: simple score, complex score, or average score. The simple score is the sum of the ratings for each question. The complex score is the sum of the ratings multiplied by a weight factor. The average score is the mean of the ratings for each domain.
Diagnostic and Statistical Manual (DSM)-5 Cross Cutting Symptom Measure | Baseline
  Students only: The DSM-5 Self-Rated Level 1 Cross-Cutting Symptom Measure-Adult is a tool designed to assess mental health domains that are important across various psychiatric diagnoses. It consists of 23 questions that evaluate 13 psychiatric domains, such as depression, anxiety, somatic symptoms, and more. Each item on the measure is rated on a 5-point scale (0=none or not at all; 1=slight or rare, less than a day or two; 2=mild or several days; 3=moderate or more than half the days; and 4=severe or nearly every day). A mild (i.e., 2) or greater rating on any item within a domain may guide additional inquiry and follow-up to determine if a more detailed assessment for that domain is necessary. Consistently high scores on a particular domain may indicate significant and problematic symptoms for the individual that might warrant further assessment, treatment, and follow-up
Students' Proactive Bystander Behavior Scale | Baseline, every 6 months up to 30 months
  This scale asks respondents to indicate whether and how often they completed proactive bystander behavior actions in the last 6 months (the time between each survey wave). Behaviors include "I have encouraged others to learn more and get involved in preventing sexual or dating violence," and "I have told guys not to talk about women in sexually degrading ways," and response options for each statement are (0) No, I have not done this in the last 6 months, (1) Yes, once in the last 6 months, and (2) Yes, more than once in the last 6 months.
Students' Reactive Bystander Action Scale | Baseline, every 6 months up to 30 months
  This scale asks respondents whether and how often they completed reactive bystander behavior actions in the last 6 months (the time between each survey wave). Actions include "I have expressed concern or offered help to a woman who said she had an unwanted sexual experience but didn't call it 'rape'," "I have reported formally to an authority a guy who used physical force against a women," and "I have intervened with a guy's action because I wanted to stop an act of sexual violence." Responses options for each statement are (0) I experienced this situation in the last 6 months and did NOT act, (1) Yes, once in the last 6 months, (2) Yes, more than once in the last 6 months, and (9) I did NOT experience any situation like this in the last 6 months.

CONTACTS AND LOCATIONS:
Overall Officials: Kathryn Yount, PhD, Principal Investigator — Emory University
Locations (7):
- Vietnam (7):
  - Can Tho University of Medicine and Pharmacy (CTUMP), Can Tho
  - Da Nang University of Medical Technology & Pharmacy (DUMTP), Da Nang
  - Hai Phong University of Medicine and Pharmacy, Haiphong
  - Hanoi Medical University, Hanoi
  - Ho Chi Minh City Medicine and Pharmacy University, Ho Chi Minh City
  - Hong Bang University, Ho Chi Minh City
  - Hue University of Medicine and Pharmacy, Huế

IPD SHARING:
Plan to Share IPD: Yes
The research team will share three waves of fully deidentified panel data with faculty; and 10 waves of fully deidentified panel data with students.
Supporting Information: Study Protocol, Analytic Code
Time Frame: Data will be made available for sharing beginning 12 months after the publication of the primary aims papers or 12 months after the end of the performance period, whichever comes first.
Access Criteria: Emory Dataverse for publicly available data and by reasonable request to the PI for any restricted data.

REFERENCES:
- [Derived] Yount KM, Whitaker D, Fang X, Trang QT, Macaulay M, Hung MT. Strategies for Implementing GlobalConsent to Prevent Sexual Violence in University Men (SCALE): Study Protocol for a National Implementation Trial. Res Sq [Preprint]. 2024 Sep 10:rs.3.rs-4745916. doi: 10.21203/rs.3.rs-4745916/v1. PMID 39315253
- [Derived] Yount KM, Whitaker DJ, Fang X, Trang QT, Macaulay M, Minh TH. Strategies for Implementing GlobalConsent to Prevent Sexual Violence in University Men (SCALE): study protocol for a national implementation trial. Trials. 2024 Aug 29;25(1):571. doi: 10.1186/s13063-024-08401-5. PMID 39210388